CLINICAL TRIAL: NCT06272968
Title: Predicting Cognition After DBS for Parkinson's Disease 2
Status: Active, not recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Dorothee Kübler, Principal Investigator, Senior Physician, Charite University, Berlin, Germany
Other Study IDs: EA2/252/23
Record Dates: First submitted 2024-02-16; First posted 2024-02-22 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Cognitive Impairment
Keywords: Cognitive Impairment; Parkinson's disease; Deep Brain Stimulation; Postoperative Delirium
MeSH Terms: conditions — Cognitive Dysfunction; Parkinson Disease; Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Neuropsychological Testing — Neuropsychological Testing via Cambridge CANTAB Connect

SUMMARY:
The aim of the study is to improve estimation of cognitive outcome after STN-DBS in PD in order to avoid risk factors by optimizing peri- and intraoperative management personalize therapeutic strategies for optimal long-term benefit.

The investigators will test possible predictors (clinical, neuropsychological, neuroimaging, electrophysiological and molecular) for the risk of cognitive dysfunction after deep brain stimulation of the subthalamic nucleus (STN-DBS) in Parkinson's disease (PD) at a single center (Charité - Universitätsmedizin Berlin, Germany). Data collection takes place prior to as well as 3, 12 and 60 months after the STN-DBS operation. Participation is proposed to all PD patients that are planned to undergo STN-DBS after careful examination of eligibility for this treatment according to standard operation procedures.

DETAILED DESCRIPTION:
Additionally to clinical routine tests, the following possible predictors of cognitive dysfunction after STN-DBS in PD are investigated:

* Imaging biomarkers: volume of the nucleus basalis of Meynert (NBM) measured on preoperative MRI and data driven search for unknown MRI characteristics relating to the incidence of postoperative neurocognitive disorder by means of Deep Learning (Convolutional Neural Networks), test of previously established classification models
* Imaging neuronal glucose metabolism with [18F]-DG PET
* Comorbidity: according to the Charlson Comorbidity Index
* Nutritional Status: defined by the Mini Nutritional Assessment (MNA-SF)
* Functional assessment of neuronal activity by 64-channel-EEG
* Duration of intra-/perioperative brake of dopaminergic medication
* Nature and depth of anaesthesia: general or conscious sedation and depth of consciousness: as measured by 4 channel electroencephalography (SedLine®) and during implantation of impulse generator
* Incidence and duration of postoperative delirium: defined according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) and/or as ≥ 2 points in the nursing Delirium Screening Scale (Nu-DESC) and/or a positive Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) score, assessment three times daily during hospital stay
* Length of stay at ICU / hospital
* Postoperative organ complications: according to Clavien-Dindo classification Localisation of bilateral electrodes and active contacts on postoperative imaging

Substudies

Correlation of domain specific CANTAB connect test scores with possible predictors and incidence of postoperative neurocognitive disorder

The resulting multivariate risk model is expected

* to improve peri- and intraoperative management by identifying avoidable risk factors for the development of postoperative cognitive deficit
* to support evidence-based and personalized decision-making when advising PD patients considering STN-DBS
* to result in the development of future hypothesis-driven interventional trials on the basis of biomarker-based sub-grouping of patients
* to allow a better understanding of underlying pathophysiological processes both PD and surgery-related regarding cognitive effects of STN-DBS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's Disease
* Indication for STN-DBS

Exclusion Criteria:

* Internistic, surgical or psychiatric contrainidications with respect to the DBS operation or treatment for the STN-DBS group
* Dementia
* Relevant language barrier

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: PD patients that are planned to undergo STN-DBS.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive performance after STN-DBS | Difference between baseline, 12 and 60 months postoperative testing
  Based on cognitive screening by Cambridge CANTAB Connect
Incidence of postoperative neurocognitive disorder | Difference between baseline, 12 and 60 months postoperative testing
  Based on cognitive screening by paper pencil test (MoCA or MDRS)

SECONDARY OUTCOMES:
Validation of post-hoc model from prior study (NCT03982953) | 1 year after DBS surgery
  MoCA1yFU = 0.7 × MoCAbaseline + 1.7 × backward spanbaseline - 1, (see https://doi.org/10.1038/s41531-025-01128-3)

CONTACTS AND LOCATIONS:
Overall Officials: Dorothee Kübler-Weller, MD, Study Chair — Movement Disorders and Neuromodulation
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided